CLINICAL TRIAL: NCT00990470
Title: Endoscopic Evaluation in Transplantation Candidates - Frequency and Prognostic Relevance of Upper and Lower Gastrointestinal Tract Findings
Brief Title: Endoscopic Evaluation in Transplantation Candidates
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Tobias J. Weismueller, Dr. T. Weismüller, Hannover Medical School
Other Study IDs: MHH-Endo-1009
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Liver Transplantation
Keywords: Transplantation; Liver; Endoscopy; Colonoscopy; Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In consideration of the limited supply of donor organs, the careful selection of transplant candidates is essential to optimize patient outcome after transplantation. Therefore an extensive evaluation of transplant candidates including among others esophagogastroduodenoscopy (EGD) and colonoscopy has been implemented in our centre. The data regarding the prevalence of upper and lower gastrointestinal (GI) pathology in transplant candidates are contradictory and are based on only a few retrospective studies, which often include only a subgroup of transplant candidates. The goal of this project is a prospective evaluation of the frequency of GI pathologies in transplant candidates with specific focus on the following questions:

1. Are there GI-pathologies that occur at a higher prevalence in transplant candidates than described in the general population and is there an increase of GI-pathologies since the introduction of the urgency-based organ allocation leading to sicker transplant candidates?
2. What is the influence of endoscopic findings on patient management before transplantation?
3. Which risk factors can be identified that predict the presence of GI-lesions?
4. Is there a subgroup of patients, in which screening colonoscopy before liver transplantation can not be recommended considering the cost/benefit ratio?
5. Is there a correlation of endoscopic findings with outcome after liver transplantation or with gastrointestinal complications during or after transplantation (e.g. gastrointestinal bleeding, perforation or gastrointestinal malignancy)?

DETAILED DESCRIPTION:
Background:

The introduction of a MELD (model for end-stage liver disease) based necessity-oriented allocation system for liver transplantation (OLT) has lead to an increasing number of patients with advanced liver disease on the waiting list. Hence it is essential to optimize outcome after transplantation in this high-risk patient collective in order to best utilize the limited supply of donor organs. To achieve this goal, the careful selection of appropriate transplantation candidates is based on an extensive evaluation of the patients including cardiac, pulmonary and renal testing and different imaging methods to exclude malignancies or an infective focus. As in many other institutions also in the Medical School Hannover (MHH) esophagogastroduodenoscopy (EGD) and colonoscopy are standard procedures during evaluation for liver transplantation. The rationale to perform these procedures is to identify patients with medical conditions that might limit their outcome after OLT. Some endoscopic findings as for example esophageal varices, gastric or duodenal ulcer or colon adenoma can be treated before transplantation, so that the patient enters the waiting list in a better medical condition. If gastrointestinal malignancies are detected, the patient will no longer be considered a candidate for OLT, unless curative treated. The detection of premalignant changes (high grade adenomas, barrett's esophagus etc.) is of great importance, since the immunosuppressed liver transplantation recipients are probably at a higher risk to progress to malignancy.

So far the data regarding the prevalence of upper and lower gastrointestinal pathologies in transplantation candidates are contradictory and are based on only a few retrospective studies. These studies often include only a subgroup of transplantation candidates. Many centres perform screening colonoscopy during OLT evaluation only in patients greater than age 45 or 50, although until today there is no clear evidence, that younger patients do not have a benefit from screening colonoscopy.

So far it is not known if certain preoperative endoscopic findings correlate with postoperative gastrointestinal complications. Such a correlation, e.g. between diverticulosis and postoperative colon perforation or peritonitis due to diverticulitis, could be highly relevant for patient management before and after OLT.

Methods:

After signing informed consent the results of EGD and colonoscopy of all patients evaluated for OLT at the MHH together with laboratory and clinical data will be entered in a database. After follow up for at least one year these data will be analyzed. Descriptive statistics as well as a multivariate analysis will be performed, to find out the frequency of endoscopic diagnoses in transplantation candidates and to look for correlations between these findings and patient outcome after OLT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive upper and/or lower endoscopy during evaluation for transplantation

Exclusion Criteria:

* patient already on waiting list

Ages: 1 Day to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients evaluated for Tranplantation at Hannover Medical School
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Wedemeyer, MD, Principal Investigator — MHH
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Derived] Weismuller TJ, Bleich F, Negm AA, Schneider A, Lankisch TO, Manns MP, Strassburg CP, Wedemeyer J. Screening colonoscopy in liver transplant candidates: risks and findings. Clin Transplant. 2013 Mar-Apr;27(2):E161-8. doi: 10.1111/ctr.12083. Epub 2013 Feb 6. PMID 23383749